CLINICAL TRIAL: NCT00960232
Title: Vitamin D, Blood Pressure, Lipids, Infection and Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UIT-ENDO-2009-1
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Hypovitaminosis D
Keywords: vitamin D; blood pressure; lipids; infection; depression
MeSH Terms: conditions — Vitamin D Deficiency; Infections; Depression | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): vitamin D 40.000 IU per weel
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Cholecalciferol — 40.000 IU cholecalciferol per week for 6 months
  Other Names: Decristol
  Arms: Vitamin D
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
There are numerous indications for a relation between low serum levels of 25(OH)D and blood pressure, lipid levels, frequency of infections and tendency towards depression. Whether it is a causal relationship it is not known, and can best be studied with a vitamin D intervention. The investigators hypothesis is that supplementation with a high dose vitamin D (40.000 IU per week) will have a beneficial effect on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* men and women 30 - 75 years of age
* low serum 25(OH)D levels

Exclusion Criteria:

* diabetes
* other serious diseases
* hypercalcemia

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Depression score | 6 months
Blood pressure | 6 months
Lipid profile | 6 months
Frequency of infections | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Jorde, Professor, Principal Investigator — University of Tromso
Locations (1):
- University of Tromsø, Tromsø, Tromsø, Norway

REFERENCES:
- [Derived] Kjaergaard M, Waterloo K, Wang CE, Almas B, Figenschau Y, Hutchinson MS, Svartberg J, Jorde R. Effect of vitamin D supplement on depression scores in people with low levels of serum 25-hydroxyvitamin D: nested case-control study and randomised clinical trial. Br J Psychiatry. 2012 Nov;201(5):360-8. doi: 10.1192/bjp.bp.111.104349. Epub 2012 Jul 12. PMID 22790678